CLINICAL TRIAL: NCT04296838
Title: Effectiveness of Conbercept in Treating Refractory Uveitic Macular Edema and the Changes of VEGF Levels in the Aqueous Humor
Brief Title: Effects of Conbercept in Refractory Uveitic Macular Edema and VEGF
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to inter-city travel restrictions for COVID-19, regular follow-up for most patients is not possible
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Bethune public welfare fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJ-LM2018010J
Record Dates: First submitted 2020-01-01; First posted 2020-03-05 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Uveitis; Macular Edema; Vascular Endothelial Growth Factor; Effect of Drugs
Keywords: Uveitis; Macular Edema; vascular endothelial growth factor; aqueous humor; Effect of Drugs
MeSH Terms: conditions — Uveitis; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- refractory UME patients treated with Conbercept (Experimental): patients in this arm should meet the inclusion criteria and the definition of refractory UME
  Interventions: Drug: intravitreal injection of Conbercept

INTERVENTIONS:
Drug: intravitreal injection of Conbercept — patients will receive intravitreal injection of Conbercept, and at the same time, aqueous humor sample will be obtained from the anterior chamber to measure the concentrations of cytokines.
  Other Names: Lumitin

SUMMARY:
As a primary exploratory study, this study aims to evaluate the short-term effectiveness of intravitreal Conbercept injection in UME, and to explore the correlation between inflammatory factors like VEGF and the responsiveness to treatment.

DETAILED DESCRIPTION:
Uveitic macular edema (UME) is one of the commonest and severest complications of chronic uveitis, and is also one of the important causes of permanent vision loss in uveitis. The pathophysiological mechanism of UME remains unclear, but was thought to be caused by damages of internal/external blood-retinal barrier mediated by inflammatory factors, including interleukin-2, interleukin-10, tumor necrosis factor α, prostaglandins and vascular endothelial growth factor (VEGF). Current treatments of UME include local or systemic glucocorticosteroids (GCS), immunosuppressants and biological agents. Although large dose of systemic GCS combined with immunosuppressants lead to quick resolution of ME in most of the cases, UME often relapse with tapering of GCS, and the side effects can be significant. Periocular or intraocular injection of GCS is effective in short term, but repetitive injections often lead to high intraocular pressure and cataract. Intravitreal injection of anti-VEGF agents is a huge advance of medical treatment in ophthalmology in recent years. Since 2007 till now, there have been a number of reports on the effectiveness of intraocular Bevacizumab and Ranibizumab injection in UME, but none about Conbercept. Besides, as the target of anti-VEGF agents, intraocular concentration of VEGF and its changes might be correlated to the sensitivity and responsiveness of UME to anti-VEGF agents, but has not been monitored. As a primary exploratory study, this study aims to evaluate the short-term effectiveness of intravitreal Conbercept injection in UME, and to explore the correlation between inflammatory factors like VEGF and the responsiveness to treatment.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years old
* competent in signing the informed consent
* no severe systemic diseases unrelated to uveitis
* fulfill the criteria of refractory UME

Exclusion Criteria:

* pregnant or preparing pregnancy
* already in other clinical trials
* blood pressure >= 180/110mmHg
* BCVA of the contralateral eye <= 20/200
* cardiovascular events within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Changes of best corrected visual acuity (BCVA) | baseline and at 1, 2, 3, 4, 5, 6 months after injection
  changes from baseline BCVA at 1, 2, 3, 4, 5, 6 months after injection (at each follow-up visit)
Changes of central retinal thickness (CRT) | baseline and at 1, 2, 3, 4, 5, 6 months after injection
  changes from baseline CRT at 1, 2, 3, 4, 5, 6 months after injection (at each follow-up visit)

SECONDARY OUTCOMES:
changes of concentration of inflammatory cytokines | before injection (baseline), 1 month after the first injection, at the end of the study (6 months)
  inflammatory cytokines include VEGF-A, VEGF-B, interleukin (IL)-2, interleukin-6, interleukin-8, interleukin-10, interleukin-12, tumor necrosis factor (TNF) α, monocyte chemotactic protein-1 and macrophage inflammatory protein-1
inflammatory status | baseline and at 1, 2, 3, 4, 5, 6 months after injection
  changes from baseline flare and cells in the anterior chamber at 1, 2, 3, 4, 5, 6 months after injection
side effects of the eye: increase of intraocular pressure | baseline and at 1, 2, 3, 4, 5, 6 months after injection
  changes from baseline intraocular pressure at 1, 2, 3, 4, 5, 6 months after injection
side effects of the eye: development/exacerbation of cataract | baseline and at 1, 2, 3, 4, 5, 6 months after injection
  whether cataract is developed or exacerbated

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital (PUMCH), Beijing, Beijing Municipality, China